CLINICAL TRIAL: NCT06769425
Title: A Phase I Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Efficacy of HS-10502 Combination Treatment in Subjects With Advanced Solid Tumors
Brief Title: HS-10502 Combination Treatment in Patients With Advanced Solid Tumors
Acronym: HS-10502
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu Hansoh Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HS-10502-103
Record Dates: First submitted 2025-01-07; First posted 2025-01-10 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Recurrent Ovarian Cancer; HER2-negative; Advanced Breast Cancer; TNBC; Advanced Prostate Cancer; Advanced Gastric Cancer
Keywords: Poly(ADP-ribose) polymerase-1 inhibitor; HS-10502; ovarian cancer; breast cancer; TNBC; prostate cancer; gastric cancer
MeSH Terms: conditions — Ovarian Neoplasms; Breast Neoplasms; Prostatic Neoplasms; Stomach Neoplasms | interventions — Platinum; Bevacizumab; 130-nm albumin-bound paclitaxel; Docetaxel; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Cohort 1 (Experimental): Advanced prostate cancer
  Interventions: Drug: HS-10502 + NHA
- Cohort 2 (Experimental): Advanced prostate cancer or solid tumor
  Interventions: Drug: HS-10502 + HS-20093
- Cohort 3 (Experimental): Advanced HER2-negative breast cancer or recurrent ovarian cancer
  Interventions: Drug: HS-10502+ Apatinib
- Cohort 4 (Experimental): Recurrent ovarian cancer
  Interventions: Drug: HS-10502 + HS-20089
- Cohort 5 (Experimental): Platinum-sensitive recurrent ovarian cancer
  Interventions: Drug: HS-10502 + Platinum + Bevacizumab
- Cohort 6 (Experimental): Advanced gastric cancer or solid tumor
  Interventions: Drug: HS-10502 + nab-paclitaxel or Docetaxel or Irinotecan
- Cohort 7 (Experimental): HRD positive advanced ovarian cancer, fallopian tube cancer or primary peritoneal cancer
  Interventions: Drug: HS-10502 + Bevacizumab

INTERVENTIONS:
Drug: HS-10502 + NHA — HS-10502 + NHA
  Arms: Cohort 1
Drug: HS-10502 + HS-20093 — HS-10502 + HS-20093
  Arms: Cohort 2
Drug: HS-10502+ Apatinib — HS-10502+ Apatinib
  Arms: Cohort 3
Drug: HS-10502 + HS-20089 — HS-10502 + HS-20089
  Arms: Cohort 4
Drug: HS-10502 + Platinum + Bevacizumab — HS-10502 + Platinum + Bevacizumab
  Arms: Cohort 5
Drug: HS-10502 + nab-paclitaxel or Docetaxel or Irinotecan — HS-10502 + nab-paclitaxel or Docetaxel or Irinotecan
  Arms: Cohort 6
Drug: HS-10502 + Bevacizumab — HS-10502 + Bevacizumab
  Arms: Cohort 7

SUMMARY:
HS-10502 is a PARP1-specific selective inhibitor. The purpose if this study is to assess the safety, tolerability, pharmacokinetics (PK), and efficacy of HS-10502 Combination Treatment in subjects with advanced solid tumors.

DETAILED DESCRIPTION:
This is a phase I, multicenter, open-label clinical study to evaluate the safety, tolerability, PK, and efficacy of oral HS-10502 combination treatment in subjects with advanced solid tumors. The study will be divided into phase Ia (dose escalation) and phase Ib (dose expansion). The dose-escalation study will be conducted to evaluate the safety, tolerability, PK profile, and efficacy, as well as to determine the maximum tolerable dosage (MTD) or maximum applicable dose (MAD) of HS-10502 in combination with other antitumor agents (Enzalutamide, Rezvilutamide,Abiraterone,HS-20093,Apatinib,HS-20089,Platinum,Bevacizumab,nab-paclitaxel,Docetaxel, Irinotecan) The subsequent dose expansion study will select appropriate target populations (7 cohorts of recurrent ovarian cancer, HER2-negative advanced breast cancer, TNBC, advanced prostate cancer , advanced gastric cancer and HRD positive advanced ovarian cancer, fallopian tube cancer or primary peritoneal cancer) based on the data obtained in the phase Ia study, and determine the recommended phase II dose (RP2D) for each target population.

Safety evaluation will be performed for all the subjects in each cycle of therapy (3 weeks or 2 weeks) until Cycle 16, and then once every 6 weeks, until 30 days or 90 days after the last dose. The PK characteristics of HS-10502 will be evaluated during screening period and study treatment. Efficacy evaluation will be performed once every 6 weeks after C1D1 until objective disease progression or withdrawal from the study. As the disease progresses, survival follow-up will be performed every 12 weeks from the last dose.

ELIGIBILITY:
Inclusion Criteria:

* Males or females aged 18 years or older (≥18 years).
* Patients diagnosed with pathologically confirmed advanced solid tumors.
* Subjects have at least one target lesion as assessed per the RECIST 1.1.
* Eastern Cooperative Oncology Group Performance Status (ECOG PS) score of 0 to 1 and no deterioration within 2 weeks before the first dose.
* Have a life expectancy of at least 12 weeks.
* Female subjects of childbearing potential are willing to take appropriate contraceptive measures and should not breastfeed from signing the informed consent until 6 months after the last dose; male subjects must agree to use barrier contraception (i.e. condoms) from signing the informed consent to 6 months after the last dose.
* Female subjects must have a negative pregnancy test within 7 days prior to the first dose (for subjects with tumor related abnormal elevation of human chorionic gonadotropin [HCG], an ultrasound of uterus and appendages should be performed within 7 days prior to the first dose to rule out pregnancy), or demonstrate no risk for pregnancy.
* Subject must be voluntarily enrolled in this clinical trial, be able to understand the study procedures and to sign written informed consent.

Exclusion Criteria:

* Have received or is currently receiving the following treatment: PARPi/B7-H4/B7-H3-targeted therapies;
* Have received or is currently receiving the following treatment: PARPi/B7-H4/B7-H3-targeted therapies;
* Have received any of cytotoxic chemotherapy drugs, investigational drugs, anti-tumor traditional Chinese medicines or other anti-tumor drugs within 14 days prior to the first dose of study drug; or need to continue these drugs during the study.
* Presence of Grade ≥ 2 toxicities as per Common Terminology Criteria for Adverse Events due to prior anti-tumor therapy.
* Presence of pleural/abdominal effusion requiring clinical intervention.
* Known history of other primary malignancy.
* Evidence of brain metastasis and/or cancerous meningitis
* Inadequate bone marrow reserve or hepatic/renal functions.
* Cardiological examination abnormality.
* Severe, uncontrolled or active cardiovascular disorders.
* Serious or poorly controlled diabetes.
* Serious or poorly controlled hypertension.
* Clinically significant bleeding symptoms or significant bleeding tendency within 1 month prior to the first dose of study treatment.
* Serious infections within 4 weeks prior to the first dose.
* Have received systemic glucocorticoid therapy for more than 7 days within 28 days prior to the first dose study treatment, or require chronic (≥ 7 days) use of systemic glucocorticoids during the study, or have other acquired, congenital immunodeficiency disorders, or a history of organ transplantation.
* Presence of active infectious diseases such as hepatitis B, hepatitis C, tuberculosis, syphilis, or human immunodeficiency virus infection, etc.
* Current hepatic encephalopathy, hepatorenal syndrome, or Child-Pugh Class B or more severe cirrhosis.
* Any moderate or severe lung diseases that may interfere with the detection and treatment of drug-related pulmonary toxicity or may seriously affect respiratory function.
* History of severe neurological or psychiatric disorder.
* Pregnant or breast-feeding women or women who intend to become pregnant during the study.
* Attenuated live vaccination within 4 weeks prior to the first dose.
* Subjects with autoimmune disease that is active or is likely to recur.
* Subjects with gastrointestinal fistula, visceral fistula, gastrointestinal perforation, or abdominal abscess, or with symptoms/signs of intestinal obstruction within 6 months prior to the first dose of study drug.
* Subjects unlikely to comply with study procedures, restrictions and requirement as determined by the investigator.
* Subjects with any condition that jeopardizes the safety of the patient or interferes with the assessment of the study, as judged by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 157 (Estimated)
Dates: Start 2025-05-07 (Actual); Primary Completion 2026-05-07 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of HS-10502（Stage 1：Dose escalating stage） | Cycle 1 (21 days)
  MTD is defined as the previous dose level at which 2 or more out of 2-6 subjects experienced a DLT.
Maximum applicable dose (MAD) of HS-10502（Stage 1：Dose escalating stage） | Cycle 1 (21days)
  MAD is defined as follows: a) based on PK data, it is anticipated that at this dose level, the dose-exposure plateau has been reached, b) based on existing safety data, it is judged that dose escalation following this dose level will have a large safety risk or subject intolerance, or c) based on the PK-PD model, it suggested that the optimal target concentration of safety and efficacy has been explored.
Efficacy of HS-10502: Objective response rate (ORR)（Stage 2： Dose expansion stage） | From the date of first dose until the date of disease progression or withdrawal from study, approximately 2 years
  ORR is defined as the proportion of participants with BOR of confirmed CR or confirmed PR per RECIST v1.1 (applicable for all solid tumors except prostate cancer) or per RECIST v1.1 and PCWG3 (for prostate cancer only).

SECONDARY OUTCOMES:
Incidence and severity of treatment-emergent adverse events | From Cycle 1 Day 1 (C1D1) until 21 days after the final dose. A cycle is 21days.
  Assessed by number and severity of adverse events as evaluated according to NCI CTCAE v5.0.
PK parameters: The maximum observed concentration (Cmax) of HS-10502 | Cycle 1 Day 1 (each cycle is 21 days)
  Defines as the maximum plasma drug concentration of HS-10502
PK parameters: time to Cmax (Tmax) of HS-10502 | Cycle 1 Day 1 (each cycle is 21 days)
  Time of maximum observed concentration of HS-10502.
PK parameters: area under the concentration-time curve from time 0 to time t of last measurable concentration (AUC0-t) of HS-10502. | Cycle 1 Day 1 (each cycle is 21 days)
  Area under the curve from the time of dosing to the time of the last measurable (positive) concentration.
PK parameters: Maximum plasma concentration at steady state (Css, max) of HS-10502 | Cycle 2 Day 1 (each cycle is 21 days)
  Defines as the maximum plasma drug concentration at steady state of HS-10502.
PK parameters: time to Css, max (Tss, max) of HS-10502 | Cycle 2 Day 1 (each cycle is 21 days)
  Time of maximum observed concentration at steady state of HS-10502.
PK parameters: Minimum plasma concentration at steady state (Css, min) of HS-10502 | Cycle 2 Day 1 (each cycle is 21 days)
  Minimum plasma drug concentration at steady state of HS-10502.
PK parameters: Area under the plasma concentration-time curve over a dosing interval at steady state (AUCss) of HS-10502 | Cycle 2 Day 1 (each cycle is 21days)
  The partial area from dosing time to dosing time plus dosing interval of HS-10502.
Efficacy of HS-10502: ORR | From the date of first dose until the date of disease progression or withdrawal from study, approximately 2 years
  ORR is defined as the proportion of participants with BOR of confirmed CR or confirmed PR per RECIST v1.1 (applicable for all solid tumors except prostate cancer) or per RECIST v1.1 and PCWG3 (for prostate cancer only).
Efficacy of HS-10502: disease control rate (DCR) | From the date of first dose until the date of disease progression or withdrawal from study, approximately 2 years
  The disease control was deﬁned as the percentage of patients who have a best overall response (confirmed CR, PR, or stable disease for at least 5 weeks) per RECIST v1.1 (applicable for all solid tumors except prostate cancer) or per RECIST v1.1 and PCWG3 (for prostate cancer only).
Efficacy of HS-10502: duration of response (DoR) | From the date of CR, PR until the date of disease progression or withdrawal from study, approximately 2 years
  DoR only applies to participants whose best overall response is CR or PR based on assessment per RECIST v1.1 (applicable for all solid tumors except prostate cancer) or per RECIST v1.1 and PCWG3 (for prostate cancer only). The start date is the date of first documented response of CR or PR (i.e. the start date of observed response, not the date when response was confirmed), and the end date is defined as the date of the first documented progression or death due to underlying cancer.
Efficacy of HS-10502: progression free survival (PFS) (applicable for all solid tumors except prostate cancer) | From the date of randomization or first dose (if randomization is not needed) until the date of disease progression or withdrawal from study, approximately 2 years.
  PFS is defined as the time from the date of randomization or first dose (if randomization is not needed) to the date of the first documented progression or death due to any cause. PFS will be assessed per RECIST v1.1.
Efficacy of HS-10502: radiographic progression free survival (rPFS) (for prostate cancer only) | From the date of randomization or first dose (if randomization is not needed) until the date of disease progression or withdrawal from study, approximately 2 years.
  rPFS is defined as the time from the date of randomization or first dose (if randomization is not needed) to the date of the first documented progression or death due to any cause. rPFS will be assessed per RECIST v1.1 (soft tissue) and PCWG3 (bone).
Efficacy of HS-10502: ORR evaluated by RECIST v1.1 and GCIG CA-125 (for ovarian cancer only) | From the date of first dose until the date of disease progression or withdrawal from study, approximately 2 years
  For ovarian cancer, ORR is defined as the proportion of participants with BOR of confirmed CR or confirmed PR per both RECIST v1.1 and GCIG CA-125 criteria.
Efficacy of HS-10502: overall survival (OS) | From the date of randomization or first dose (if randomization is not needed) until the documentation of death from any cause, approximately 4 years
  OS is defined as the time from the date of randomization or first dose (if randomization is not needed) to the date of death due to any cause. For each participant who is not known to have died as of the cutoff date for overall survival analysis, OS time was censored on the last date the participant is known to be alive.
Efficacy of HS-10502: Proportion of subjects with CA-125 decreased by ≥ 50% from baseline (for ovarian cancer only) | From the date of first dose until the date of disease progression or withdrawal from study, approximately 2 years
  The percentage of subjects (ovarian cancer only) with a reduction of at least 50% from baseline in CA-125 levels.
Efficacy of HS-10502: PSA50 response rate (for prostate cancer only) | From the date of first dose until the date of disease progression or withdrawal from study, approximately 2 years
  PSA50 response rate is defined as the proportion of subjects with a PSA nadir of ≤ 50% of baseline PSA level confirmed by serial PSA assessments (at least 3 weeks apart) after the start of the study.
Efficacy of HS-10502: Time to PSA progression (for prostate cancer only) | From the date of first dose until the date of disease progression or withdrawal from study, approximately 2 years
  Time to PSA progression is defined as the time from the first dose to PSA progression based on PCWG3 criteria.

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No